CLINICAL TRIAL: NCT03737383
Title: Treating Violence-related PTSD and Substance Risk in Low-income, Urban Adolescents
Acronym: POWER-NET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Jennifer Read, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00000298; UL1TR001412 (NIH)
Record Dates: First submitted 2018-01-29; First posted 2018-11-09 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Posttraumatic Stress Disorder; Substance Use Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility and Preliminary Efficacy (Experimental): We will be administering Narrative Exposure Therapy to determine participant responses to the intervention, whether the intervention can be delivered successfully in this setting, and preliminary outcomes.
  Interventions: Behavioral: Narrative Exposure Therapy

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — brief, trauma-focused treatment.
  Other Names: NET

SUMMARY:
This project will provide initial feasibility and efficacy data for the implementation of Narrative Exposure Therapy (NET) to urban, at-risk youth. Posttraumatic stress and substance use outcomes, as well as participant responses to the intervention, will be examined.

DETAILED DESCRIPTION:
The goal of the proposed study is to gather preliminary feasibility and efficacy data for an innovative intervention (Narrative Exposure Therapy: NET) to promote adolescent mental health related to interpersonal trauma (IPT). Among those at highest risk for interpersonal violence and its sequelae are youth from urban, low-resourced neighborhoods. Post-traumatic stress disorder (PTSD) is a common outcome associated with IPT. Substance misuse (SUB) is a frequent concomitant of PTSD. NET is a promising intervention to reduce PTSD symptoms and associated psychological distress, via the supported reconstruction (narrative telling) of the traumas. NET has a critical advantage over existing PTSD treatments in that it can be delivered in a brief format, in community settings where at-risk adolescents are likely to be found. Despite its promise in treating adolescent distress, NET has yet to be tested as an intervention for those who have interpersonal trauma-related PTSD. Further NET's influence on SUB has not been examined.

Accordingly, the objective of this project is to conduct a pilot study (N=30) to estimate NET treatment effects on PTSD symptoms and SUB in IPT-exposed urban adolescents (ages 16-21). Both feasibility and preliminary efficacy data will be collected to serve as pilot work for a larger-scale NIH proposal. Recruitment and intervention will be set within community partners where the adolescents already are connected and are receiving social or psychological services. Outcome data will be collected at: (T0) Baseline, and at 1(T1), and 3 months (T2) follow-up assessments. Participant responses to the intervention will be assessed post-intervention. Change in PTSD, SUB will be estimated with effect sizes and inferential tests. Preliminary evidence of efficacy and feasibility will pave the way for further NET development to offer a patient-oriented, community-based, intervention that will promote adolescent mental health for those at greatest risk for health access and outcomes disparities.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (ages 16-25),
* Positive PTSD diagnosis (CAPS diagnosis)
* Positive lifetime incidence of interpersonal violence-related trauma.

Exclusion Criteria:

* Actively suicidal with an immediate referral to the community agency crisis staff
* Severe cognitive delay
* Active psychosis

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist-Civilian Version | through study completion, an average of 3 years
  assessed via PTSD checklist. The minimum score for this measure is 0 while the maximum is 80. Higher scores indicate more severe PTSD symptoms.

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | through study completion, an average of 3 years
  alcohol use assessed via AUDIT. The minimum score for this measure is 0 while the maximum is 40. Higher scores indicate more alcohol use.
Young Adult Alcohol Consequences Questionnaire (YAACQ) | through study completion, an average of 3 years
  alcohol consequences assessed via YAACQ. The minimum score for this measure is 0 while the maximum is 48. Higher scores indicate more alcohol consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Tiffany, Ph.D., Study Chair — University at Buffalo
Locations (1):
- University at Buffalo Department of Psychology, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share a de-identified data set which will include baseline demographics and trauma, PTSD, and drinking outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available in June of 2020 and will be available until 2025.
Access Criteria: There must be an articulation of a clear research question and analytic plan by an established investigator with the relevant credentials. The information will be shared as a digital file through email.